CLINICAL TRIAL: NCT02447458
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Safety, Tolerability, and Pharmacokinetics Study of Escalating Single Doses of MLN3126 in Healthy Subjects
Brief Title: MLN3126 Single Rising Dose Study
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Site non-compliance to GCP (No safety concerns. See detailed description)
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MLN3126_102; U1111-1163-1717 (Other: Universal Trial Number (WHO))
Record Dates: First submitted 2015-05-14; First posted 2015-05-18 (Estimated); Results first posted 2015-08-05 (Estimated); Last update posted 2015-08-05 (Estimated); Status verified 2015-07

CONDITIONS: Healthy Volunteers
Keywords: Drug therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (7):
- Cohort 1: MLN3126 300 mg (Experimental): MLN3126 300 mg tablets, orally, fasting, once on Day 1.
  Interventions: Drug: MLN3126
- Cohort 2: MLN3126 600 mg (Experimental): MLN3126 600 mg tablets, orally, fasting, once on Day 1.
  Interventions: Drug: MLN3126
- Cohort 3: MLN3126 1000 mg (Experimental): MLN3126 1000 mg tablets, orally, fasting, once on Day 1. Participants returned to the clinic then received MLN3126 1000 mg tablets, orally, fed (30 minutes after the start of a high-fat breakfast), once on Day 1.
  Interventions: Drug: MLN3126
- Cohort 4: MLN3126 1500 mg (Experimental): MLN3126 1500 mg administered orally as tablets, once on Day 1.
  Interventions: Drug: MLN3126
- Cohort 5: MLN3126 2000 mg (Experimental): MLN3126 2000 mg tablets, orally, fasting, once on Day 1.
  Interventions: Drug: MLN3126
- Cohort 6 (Experimental): Did not take place due to termination of the study.
  Interventions: Drug: MLN3126
- Placebo: Cohort 1-6 (Placebo Comparator): Placebo-matching MLN3126 tablets, orally, once on Day 1.
  Interventions: Drug: MLN3126 Placebo

INTERVENTIONS:
Drug: MLN3126 — MLN3126 tablets
  Arms: Cohort 1: MLN3126 300 mg; Cohort 2: MLN3126 600 mg; Cohort 3: MLN3126 1000 mg; Cohort 4: MLN3126 1500 mg; Cohort 5: MLN3126 2000 mg; Cohort 6
Drug: MLN3126 Placebo — MLN3126 placebo-matching tablets
  Arms: Placebo: Cohort 1-6

SUMMARY:
The purpose of this study was to evaluate the safety, tolerability, and pharmacokinetics of MLN3126 when administered as a single dose of tablets at escalating dose levels in healthy participants.

DETAILED DESCRIPTION:
The drug tested in this study is called MLN3126. The study evaluated the safety, tolerability, pharmacokinetics (PK), pharmacodynamics and the potential effect of food on the PK of MLN3126 and its M-I metabolite following single oral dose administrations.

This study planned to enroll approximately 48 healthy participants, who were to be enrolled in 1 of the 6 dose cohorts or matching placebo in an ascending fashion. Participants were randomly assigned to MLN3126 or placebo within each cohort- which remained undisclosed to the participant and study doctor during the study (unless there was an urgent medical need):

* Cohort 1 - MLN3126 300 mg or matching placebo
* Cohort 2 - MLN3126 600 mg or matching placebo
* Cohort 3 - MLN3126 1000 mg or matching placebo
* Cohort 3 - MLN3126 1000 mg or matching placebo (fed regimen)
* Cohort 4 - MLN3126 1500 mg or matching placebo
* Cohort 5 - MLN3126 2000 mg or matching placebo
* Cohort 6 - Did not taken place due to termination of the study

All participants were asked to take the required tablets at the same time throughout the study.

This single-centre trial was conducted in The United States. Participants were confined to the clinic for 5 days, and were contacted by telephone on day 14 (±2days) for a follow-up assessment.

This study was terminated after completion of Cohort 5 due to findings of study site non-compliance to Good Clinical Practice (GCP) regarding study documentation. There were no safety concerns.

ELIGIBILITY:
Inclusion Criteria:

1. In the opinion of the investigator, the participant was capable of understanding and complying with protocol requirements.
2. The participant or, when applicable, the participant's legally acceptable representative signed and dated a written, informed consent form and any required privacy authorization prior to the initiation of any study procedures.
3. Is a male or female adult, aged 18 to 55 years, inclusive, at the time of informed consent and study drug dosing.
4. Is a healthy adult male or female subject as evidenced by their medical history, complete physical examination, vital signs, ECG, and safety laboratory evaluations.
5. Weighed at least 45 kg (99 lbs) and had a body mass index (BMI) between 18 and 30.0 kg/m2 inclusive at Screening.
6. A male participant who was nonsterilized and sexually active with a female partner of childbearing potential agreed to use adequate contraception from signing of informed consent throughout the duration of the study and for 12 weeks after last dose. In addition, participants were advised not to donate sperm during this period.
7. A female participant of childbearing potential who was sexually active with a nonsterilized male partner agreed to use routinely adequate contraception from signing of informed consent throughout the duration of the study to their next postconfinement menstruation. In addition participants were advised not to donate ova during this period.

Exclusion Criteria:

Any participant who meets any of the following criteria will not qualify for entry into the study:

1. Has received any investigational compound within 30 days prior to the first dose of study medication.
2. Is an immediate family member, study site employee, or in a dependent relationship with a study site employee who is involved in the conduct of this study (eg, spouse, parent, child, sibling) or may consent under duress.
3. Has uncontrolled, clinically significant neurologic, cardiovascular, pulmonary, hepatic, renal, metabolic, GI, or endocrine disease or other abnormality, which may impact the ability of the participant to participate or potentially confound the study results.
4. Has a known hypersensitivity to any component of the formulation of MLN3126.
5. Has a positive urine drug result for drugs of abuse at Screening or Check-in (Day -1).
6. Has a history of drug abuse (defined as any illicit drug use) or a history of alcohol abuse (defined as 4 alcoholic beverages per day) within 1 year prior to the Screening visit or is unwilling to agree to abstain from alcohol and drugs throughout the study.
7. Has taken any excluded medication, supplements, or food products listed in the Excluded Medications and Dietary Products section of the protocol.
8. If female, the participant is pregnant or lactating or intending to become pregnant, or intending to donate ova, before or during, the study; including the timeframe to participant's next postconfinement menstruation after participating in this study.
9. If male, the participant intends to donate sperm during the course of this study or for 12 weeks thereafter.
10. Has evidence of current cardiovascular, central nervous system, hepatic, hematopoietic disease, renal dysfunction, metabolic or endocrine dysfunction, serious allergy, asthma hypoxemia, hypertension, seizures, or allergic skin rash. There is any finding in the participant's medical history, physical examination, or safety laboratory tests giving reasonable suspicion of a disease that would contra indicate taking MLN3126 or a similar drug in the same class, or that might interfere with the conduct of the study. This includes, but is not limited to, peptic ulcer disease, seizure disorders, and cardiac arrhythmias.
11. Has current or recent (within 6 months) GI disease that would be expected to influence the absorption of drugs (ie, a history of malabsorption, any surgical intervention known to impact absorption [eg, bariatric surgery or bowel resection], esophageal reflux, peptic ulcer disease, erosive esophagitis or frequent [more than once per week] occurrence of heartburn).
12. Has a history of cancer or other malignancy, except basal cell carcinoma that has been in remission for at least 5 years prior to Day 1.
13. Has a positive test result for hepatitis B surface antigen, antibody to hepatitis C virus, at Screening or a known history of human immunodeficiency virus infection.
14. Has used nicotine-containing products (this includes, but is not limited to, cigarettes, pipes, cigars, chewing tobacco, nicotine patch or nicotine gum) within 28 days prior to Check-in Day -1. Cotinine test is positive at Screening or Check-in (Day -1).
15. Has poor peripheral venous access.
16. Has donated or lost 450 mL or more of his or her blood volume (including plasmapheresis), or had a transfusion of any blood product within 45 days prior to Day 1.
17. Has a Screening or Check-in (Day -1) abnormal (clinically significant) ECG. Entry of any subject with an abnormal (not clinically significant) ECG must be approved, and documented by signature by the principal investigator or medically qualified subinvestigator.
18. Has abnormal Screening or Check-in (Day -1) laboratory values that suggest a clinically significant underlying disease or participant with the following laboratory abnormalities: alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) >1.5×ULN.
19. Has QT interval with Fridericia correction method (QTcF) >430 ms for men and >450 ms for women or PR outside the range of 120 to 220 ms confirmed upon repeat testing within a maximum of 5 minutes, at the Screening Visit or Check-in (Day -1).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2013-09; Primary Completion 2014-01 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Eatontown, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1 investigative site in the United States from 19 August 2013 (first participant signed informed consent form) to 05 February 2014.
Pre-assignment Details: Healthy volunteers were enrolled in 1 of 5 MLN3126 ascending dose treatment groups: once a day 300 mg, 600 mg, 1000 mg under fed or fasting conditions,1500 mg or 2000 mg OR once a day placebo.
Groups:
- MLN3126 300 mg: MLN3126 300 mg tablets, orally, fasting, once on Day 1.
- MLN3126 600 mg: MLN3126 600 mg tablets, orally, fasting, once on Day 1.
- MLN3126 1000 mg: MLN3126 1000 mg tablets, orally, fasting, once on Day 1. Participants returned to the clinic then received MLN3126 1000 mg tablets, orally, fed (30 minutes after the start of a high-fat breakfast), once on Day 1.
- MLN3126 1500 mg: MLN3126 1500 mg tablets, orally, fasting, once on Day 1.
- MLN3126 2000 mg: MLN3126 2000 mg tablets, orally, fasting once on Day 1.
- Placebo: Placebo-matching MLN3126 tablets, orally, fasting, once on Day 1.
Period: Overall Study
Arm/Group | MLN3126 300 mg | MLN3126 600 mg | MLN3126 1000 mg | MLN3126 1500 mg | MLN3126 2000 mg | Placebo
Started | 5 | 6 | 6 | 6 | 6 | 10
Completed | 5 | 6 | 5 | 6 | 6 | 10
Not Completed | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MLN3126 300 mg | MLN3126 600 mg | MLN3126 1000 mg | MLN3126 1500 mg | MLN3126 2000 mg | Placebo | Total
Number analyzed (Participants) | 5 | 6 | 6 | 6 | 6 | 10 | 39
Age, Continuous [Mean (Standard Deviation); unit: Years] | 36.8 (10.43) | 30.3 (6.50) | 41.2 (10.42) | 32.3 (11.78) | 30.0 (8.39) | 32.8 (6.32) | 33.7 (9.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 2 | 3 | 1 | 3 | 15
  Male | 2 | 3 | 4 | 3 | 5 | 7 | 24
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Black or African American | 2 | 6 | 3 | 5 | 5 | 7 | 28
  White | 2 | 0 | 3 | 1 | 1 | 3 | 10
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 2 | 0 | 2 | 2 | 1 | 3 | 10
  Non-Hispanic or Latino | 3 | 6 | 4 | 4 | 5 | 7 | 29
Height [Mean (Standard Deviation); unit: cm] | 170.8 (10.64) | 172.3 (5.47) | 174.7 (10.42) | 169.8 (5.71) | 173.3 (6.09) | 174.9 (13.08) | 172.9 (9.14)
Weight [Mean (Standard Deviation); unit: kg] | 78.00 (12.900) | 81.98 (8.538) | 83.67 (15.871) | 72.22 (7.165) | 75.87 (10.016) | 82.58 (7.420) | 79.44 (10.498)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 26.65 (2.643) | 27.56 (2.127) | 27.18 (2.293) | 25.01 (1.811) | 25.16 (2.329) | 27.22 (3.251) | 26.54 (2.587)
Caffeine Consumption [Number; unit: participants]
  Yes | 1 | 1 | 2 | 3 | 0 | 3 | 10
  No | 4 | 5 | 4 | 3 | 6 | 7 | 29
Smoking Classification [Number; unit: participants]
  Never smoked | 5 | 6 | 4 | 6 | 6 | 10 | 37
  Current smoker | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Ex-smoker | 0 | 0 | 2 | 0 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Experience At Least One Treatment-Emergent Adverse Event (TEAE) Post-Dose
Description: An Adverse Event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (eg, a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug. A treatment-emergent adverse event (TEAE) is defined as an adverse event with an onset that occurs after receiving study drug.
Time Frame: Up to Day 22
Population: Safety population included all enrolled participants who received at least 1 dose of study drug.
Measure: Number; unit: Participants
Groups:
- MLN3126 1000 mg (Fed): MLN3126 1000 mg tablets, orally, fed (30 minutes after the start of a high-fat breakfast), once on Day 1.
- Placebo (Fed): Placebo matching MLN3126 tablets, orally, fed (30 minutes after the start of a high-fat breakfast), once on Day 1.
Arm/Group | MLN3126 300 mg | MLN3126 600 mg | MLN3126 1000 mg | MLN3126 1500 mg | MLN3126 2000 mg | Placebo | MLN3126 1000 mg (Fed) | Placebo (Fed)
Number analyzed (Participants) | 5 | 6 | 6 | 6 | 6 | 10 | 5 | 2
Participants | 1 | 0 | 1 | 0 | 1 | 1 | 1 | 0

2. Primary Outcome: Percentage of Participants With Markedly Abnormal Clinical Laboratory Results Post-Dose
Description: Clinical safety laboratory tests included clinical chemistry, hematology and urinalysis. The percentage of participants with any markedly abnormal laboratory finding during the study.
Time Frame: Up to Day 16
Population: Safety population included all enrolled participants who received at least 1 dose of study drug.
Measure: Number; unit: Percentage of Participants
Arm/Group | MLN3126 300 mg | MLN3126 600 mg | MLN3126 1000 mg | MLN3126 1500 mg | MLN3126 2000 mg | Placebo | MLN3126 1000 mg (Fed) | Placebo (Fed)
Number analyzed (Participants) | 5 | 6 | 6 | 6 | 6 | 10 | 5 | 2
Percentage of Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Percentage of Participants With Markedly Abnormal Vital Signs Post-Dose
Description: Vital signs included oral body temperature measurement, blood pressure, respiration rate, and pulse rate [beats per minute (bpm) or heart rate]. The percentage of participant with markedly abnormal vital signs findings during the study. OBP=Orthostatic Blood Pressure. All OBP measurements were standing.
Time Frame: Up to Day 16
Population: Safety population included all enrolled participants who received at least 1 dose of study drug.
Measure: Number; unit: Percentage of Participants
Arm/Group | MLN3126 300 mg | MLN3126 600 mg | MLN3126 1000 mg | MLN3126 1500 mg | MLN3126 2000 mg | Placebo | MLN3126 1000 mg (Fed) | Placebo (Fed)
Number analyzed (Participants) | 5 | 6 | 6 | 6 | 6 | 10 | 5 | 2
Percentage of Participants
  Pulse - supine | 0 | 33.3 | 33.3 | 16.7 | 33.3 | 40.0 | 0 | 0
  Pulse - standing 1 minute | 40.0 | 50.0 | 0 | 16.7 | 16.7 | 20.0 | 40.0 | 0
  Pulse - standing 3 minutes | 20.0 | 50.0 | 0 | 16.7 | 0 | 10.0 | 40.0 | 0
  Systolic Blood pressure (BP) - supine | 20.0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Systolic Blood pressure - standing 1 minute | 0 | 0 | 0 | 0 | 0 | 0 | 20.0 | 0
  Systolic Blood pressure - standing 3 minutes | 0 | 0 | 16.7 | 16.7 | 0 | 0 | 20.0 | 0
  Diastolic blood pressure - supine | 40.0 | 33.3 | 0 | 16.7 | 16.7 | 20.0 | 20.0 | 50.0
  Diastolic blood pressure - standing 1 minute | 20.0 | 33.3 | 33.3 | 0 | 16.7 | 30.0 | 40.0 | 50.0
  Diastolic blood pressure - standing 3 minutes | 20.0 | 0 | 0 | 16.7 | 0 | 20.0 | 40.0 | 0
  OBP systolic - 1 minutes (Decrease of >40 mmHg) | 0 | 0 | 0 | 16.7 | 0 | 0 | 0 | 0
  OBP systolic - 3 minutes (Decrease of >40 mmHg) | 0 | 0 | 0 | 16.7 | 0 | 0 | 0 | 0
  OBP diastolic - 1 minutes (Decrease >20 mmHg) | 40.0 | 0 | 33.3 | 33.3 | 33.3 | 40.0 | 20.0 | 100.0
  OBP diastolic - 3 minutes (Decrease >20 mmHg) | 0 | 16.7 | 33.3 | 50.0 | 33.3 | 50.0 | 0 | 50.0

4. Primary Outcome: Percentage of Participants With Markedly Abnormal Electrocardiogram (ECG) Findings Post-Dose
Description: A standard 12-lead ECG was performed. The percentage of participants with markedly abnormal electrocardiogram (ECG) findings during the study.
Time Frame: Up to Day 16
Population: Safety population included all enrolled participants who received at least 1 dose of study drug.
Measure: Number; unit: Percentage of Participants
Arm/Group | MLN3126 300 mg | MLN3126 600 mg | MLN3126 1000 mg | MLN3126 1500 mg | MLN3126 2000 mg | Placebo | MLN3126 1000 mg (Fed) | Placebo (Fed)
Number analyzed (Participants) | 5 | 6 | 6 | 6 | 6 | 10 | 5 | 2
Percentage of Participants
  Heart Rate | 0 | 16.7 | 0 | 16.7 | 33.3 | 20.0 | 0 | 0
  PR Interval | 0 | 16.7 | 33.3 | 0 | 33.3 | 10.0 | 40.0 | 0
  QRS Interval | 0 | 0 | 0 | 0 | 0 | 10.0 | 0 | 0
  QTc - Fredericia's | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QTc Interval | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Cmax: Maximum Plasma Concentration of MLN3126 and Metabolite M-I
Description: Maximum observed plasma concentration (Cmax) is the peak plasma concentration of a drug after administration, obtained directly from the plasma concentration-time curve.
Time Frame: Pre-dose and multiple timepoints post-dose (Up to 96 Hours)
Population: Pharmacokinetic (PK) analysis set included all participants who received study drug and who had at least 1 measurable PK plasma concentration.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | MLN3126 300 mg | MLN3126 600 mg | MLN3126 1000 mg | MLN3126 1500 mg | MLN3126 2000 mg | MLN3126 1000 mg (Fed)
Number analyzed (Participants) | 5 | 6 | 6 | 6 | 6 | 5
ng/mL
  MLN3126 | 2466.00 (387.208) | 3605.00 (920.885) | 4061.67 (1192.299) | 5490.00 (1110.531) | 8200.00 (1937.431) | 9444.00 (1929.632)
  MLN3126 M-I Metabolite | 125.26 (44.940) | 238.17 (101.275) | 278.17 (176.552) | 374.00 (78.908) | 424.83 (131.574) | 684.40 (556.234)

6. Secondary Outcome: Tmax: Time to Maximum Plasma Concentration of MLN3126 and Metabolite M-I
Description: Tmax is the time to reach the maximum plasma concentration (Cmax), equal to time (hours) to Cmax.
Time Frame: Pre-dose and multiple timepoints post-dose (Up to 96 Hours)
Population: PK analysis set included all participants who received study drug and who had at least 1 measurable PK plasma concentration.
Measure: Median (Full Range); unit: Hours
Arm/Group | MLN3126 300 mg | MLN3126 600 mg | MLN3126 1000 mg | MLN3126 1500 mg | MLN3126 2000 mg | MLN3126 1000 mg (Fed)
Number analyzed (Participants) | 5 | 6 | 6 | 6 | 6 | 5
Hours
  MLN3126 | 2.00 (1.884) [1.50 to 6.00] | 3.00 (0.894) [2.00 to 4.00] | 3.14 (0.902) [2.00 to 4.00] | 2.50 (2.345) [2.00 to 8.00] | 3.01 (0.752) [2.00 to 4.00] | 6.00 [4.00 to 10.00]
  MLN3126 M-I Metabolite | 4.00 [4.00 to 6.00] | 4.00 [4.00 to 8.00] | 4.00 [4.00 to 8.00] | 4.00 [4.00 to 10.00] | 4.00 [4.00 to 8.00] | 8.00 [6.00 to 10.00]

7. Secondary Outcome: AUC(0-tlqc): Area Under the Plasma Concentration Time Curve of MLN3126 and Metabolite M-I From Time 0 to the Last Quantifiable Concentration
Description: AUC(0-tlqc) is a measure of total plasma exposure to the drug from Time 0 to Time of the Last Quantifiable Concentration (AUC[0-tlqc]).
Time Frame: Pre-dose and multiple timepoints post-dose (Up to 96 Hours)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | MLN3126 300 mg | MLN3126 600 mg | MLN3126 1000 mg | MLN3126 1500 mg | MLN3126 2000 mg | MLN3126 1000 mg (Fed)
Number analyzed (Participants) | 5 | 6 | 6 | 6 | 6 | 5
ng*hr/mL
  MLN3126 | 41480.14 (7541.025) | 63117.71 (26292.596) | 73474.61 (29655.501) | 108475.58 (20425.152) | 133029.91 (44849.002) | 248462.35 (72106.157)
  MLN3126 M-I Metabolite | 1961.73 (1106.451) | 4096.06 (2261.405) | 5550.19 (5139.476) | 6724.92 (2067.765) | 6110.64 (1936.969) | 11989.43 (10546.217)

8. Secondary Outcome: AUC(0-inf): Area Under the Plasma Concentration Time Curve of MLN3126 and Metabolite M-I From Time 0 to Infinity
Description: AUC(0-inf) is measure of area under the curve from time 0 to infinity.
Time Frame: Pre-dose and multiple timepoints post-dose (Up to 96 Hours)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | MLN3126 300 mg | MLN3126 600 mg | MLN3126 1000 mg | MLN3126 1500 mg | MLN3126 2000 mg | MLN3126 1000 mg (Fed)
Number analyzed (Participants) | 5 | 6 | 6 | 6 | 6 | 5
ng*hr/mL
  MLN3126 | 41765.17 (7549.827) | 63508.18 (26520.426) | 78964.45 (40182.582) | 110437.12 (20911.078) | 134119.22 (45470.528) | 250789.67 (73569.482)
  MLN3126 M-I Metabolite | 1993.65 (1099.291) | 4132.89 (2266.377) | 6668.14 (7725.447) | 6949.52 (2129.918) | 6177.45 (1977.067) | 12068.75 (10609.268)

9. Secondary Outcome: CL/F: Oral Clearance of MLN3126
Description: CL/F is apparent clearance of the drug from the plasma, after extravascular administration.
Time Frame: Pre-dose and multiple timepoints post-dose (Up to 96 Hours)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: L/hr
Arm/Group | MLN3126 300 mg | MLN3126 600 mg | MLN3126 1000 mg | MLN3126 1500 mg | MLN3126 2000 mg | MLN3126 1000 mg (Fed)
Number analyzed (Participants) | 5 | 6 | 6 | 6 | 6 | 5
L/hr | 7.39 (1.457) | 11.34 (5.934) | 15.12 (6.345) | 13.97 (2.473) | 16.76 (6.656) | 4.23 (1.066)

10. Secondary Outcome: T ½: Half-life of MLN3126 and Metabolite M-I
Description: Terminal phase elimination half-life (T1/2) is the time required for half of the drug to be eliminated from the plasma.
Time Frame: Pre-dose and multiple timepoints post-dose (Up to 96 Hours)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | MLN3126 300 mg | MLN3126 600 mg | MLN3126 1000 mg | MLN3126 1500 mg | MLN3126 2000 mg | MLN3126 1000 mg (Fed)
Number analyzed (Participants) | 5 | 6 | 6 | 6 | 6 | 5
Hours
  MLN3126 | 13.94 (0.992) | 12.80 (0.624) | 16.07 (5.899) | 16.31 (3.706) | 13.63 (1.888) | 13.92 (0.894)
  MLN3126 M-I Metabolite | 13.44 (1.815) | 13.47 (1.524) | 19.88 (16.767) | 20.89 (9.006) | 14.09 (3.053) | 13.56 (1.960)

11. Secondary Outcome: Ae (0-96): Total Amount of MLN3126 and Metabolite M-I Excreted in the Urine
Description: Ae (0-96) is the total amount of drug excreted in urine from time 0 to time 96 hours.
Time Frame: Pre-dose and multiple timepoints post-dose (Up to 96 Hours)
Population: PK analysis set included all participants who received study drug and who had at least 1 measurable PK urine concentration.
Measure: Mean (Standard Deviation); unit: ng
Arm/Group | MLN3126 300 mg | MLN3126 600 mg | MLN3126 1000 mg | MLN3126 1500 mg | MLN3126 2000 mg | MLN3126 1000 mg (Fed)
Number analyzed (Participants) | 5 | 6 | 6 | 6 | 6 | 5
ng
  MLN3126 | 65864.50 (13803.378) | 128194.87 (41264.086) | 115101.67 (101342.371) | 115443.11 (45489.137) | 179199.95 (94480.203) | 216883.09 (193535.668)
  MLN3126 M-I Metabolite | 1606271.00 (661316.505) | 3785848.92 (1487530.534) | 3669719.92 (3805989.870) | 3042712.33 (1087430.529) | 4934093.92 (2367261.267) | 7969436.83 (9141564.346)

12. Secondary Outcome: Fe: Fraction of MLN3126 Excreted in the Urine
Description: Fe is the Fraction of drug excreted in urine, calculated as Fe=(Ae[0-t]/dose)×100.
Time Frame: Pre-dose and multiple timepoints post-dose (Up to 96 Hours)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | MLN3126 300 mg | MLN3126 600 mg | MLN3126 1000 mg | MLN3126 1500 mg | MLN3126 2000 mg | MLN3126 1000 mg (Fed)
Number analyzed (Participants) | 5 | 6 | 6 | 6 | 6 | 5
Percentage | 0.02 (0.005) | 0.02 (0.007) | 0.01 (0.002) | 0.01 (0.003) | 0.01 (0.005) | 0.01 (0.007)

13. Secondary Outcome: Renal Clearance (CLr) of MLN3126 and Metabolite M-I
Description: Renal clearance was calculated as CLr=Ae(0-96)/AUC (0-96).
Time Frame: Pre-dose and multiple timepoints post-dose (Up to 96 Hours)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | MLN3126 300 mg | MLN3126 600 mg | MLN3126 1000 mg | MLN3126 1500 mg | MLN3126 2000 mg | MLN3126 1000 mg (Fed)
Number analyzed (Participants) | 5 | 6 | 5 | 6 | 6 | 4
mL/min
  MLN3126 | 0.03 (0.010) | 0.04 (0.010) | 0.02 (0.010) | 0.02 (0.010) | 0.02 (0.012) | 0.01 (0.004)
  MLN3126 M-I Metabolite | 16.00 (9.945) | 16.15 (3.426) | 10.34 (7.285) | 7.89 (2.544) | 13.69 (7.728) | 9.05 (5.598)

ADVERSE EVENTS:
Time Frame: First dose of study drug to 30 days post last dose (Up to Day 31)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | MLN3126 300 mg | MLN3126 600 mg | MLN3126 1000 mg | MLN3126 1500 mg | MLN3126 2000 mg | Placebo | MLN3126 1000 mg (Fed) | Placebo (Fed)
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/6 | 0/6 | 0/6 | 0/6 | 0/10 | 0/5 | 0/2
Other Adverse Events (participants affected / at risk) | 1/5 | 0/6 | 1/6 | 0/6 | 1/6 | 1/10 | 1/5 | 0/2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MLN3126 300 mg (N=5) | MLN3126 600 mg (N=6) | MLN3126 1000 mg (N=6) | MLN3126 1500 mg (N=6) | MLN3126 2000 mg (N=6) | Placebo (N=10) | MLN3126 1000 mg (Fed) (N=5) | Placebo (Fed) (N=2)
Headache (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.